CLINICAL TRIAL: NCT02208830
Title: Effects of Pulmonary Rehabilitation Associated With Respiratory Therapy vs Physiotherapy in Physical Capacity, Peripheral Muscle Strength and Quality of Life in Patients With Bronchiectasis: a Randomized Controlled Trial.
Brief Title: Physical Capacity in Patients With Bronchiectasis Before and After Rehabilitation Program
Acronym: PCBCQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Anderson Alves de Camargo, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BCQPC
Record Dates: First submitted 2012-03-07; First posted 2014-08-05 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; functional capacity; lung functional
MeSH Terms: conditions — Bronchiectasis | interventions — Exercise; Rehabilitation; Therapeutics; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional program (Experimental): The conventional program is conducted with duration of 8 week, twice weekly. The techniques used will be: expiration with the glottis open in lateral posture (Eltgol), autogenous drainage (AD) and shaker. Each technique will last for 30 minutes.
  Interventions: Other: conventional program
- pulmonary rehabilitation (Experimental): Duration of 8 week, twice weekly exercise program with: lower limb strength training and aerobic training per 30 minutes.
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — Pulmonary rehabilitation: 8 week, twice weekly exercise program with aerobic treadmill training and lower limb strength training.
  Other Names: exercise; rehabilitation; treatment; pulmonary
  Arms: pulmonary rehabilitation
Other: conventional program — The conventional program is conducted with duration of 8 week, twice weekly. The techniques used will be: expiration with the glottis open in lateral posture (Eltgol), autogenous drainage (AD) and shaker. Each technique will last for 30 minutes.
  Other Names: physiotherapy; treatment respiratory
  Arms: conventional program

SUMMARY:
The hypothesis of this study is that the group of patients who will carry out the rehabilitation program associated with respiratory therapy will have higher benefits in physical function, peripheral muscle strength and quality of life compared to the group that will only perform chest physiotherapy. Additionally, there will be a negative correlation between inflammatory mediators and measures of physical ability as well as the magnitude of improvement is lower after treatment in patients with higher baseline levels of inflammation. Furthermore, these patients will be reevaluated in 1 and 3 years, as a cohort, studying if exercise capacity may be a predictor of clinical and functional outcomes.

DETAILED DESCRIPTION:
All patients will have their dyspnea rated according to the Medical Research Council (MRC) scale. The Saint George Respiratory Questionnaire (SGRQ) and COPD Assessment test (CAT) will also be applied.

Spirometry will be performed according to recommendations of the American Thoracic Society/European Respiratory Society. The forced vital capacity and forced expiratory volume values in the first second will be compared with those predicted for the Brazilian population.

The maximal incremental cycle ergometer test will be carried out on an electromagnetically braked cycle ergometer with gas exchange and ventilatory variables analyzed breath-by-breath. After 2 min at rest and then 2 min pedaling in freewheel, the power (W) will continuously increase in a linear "ramp" pattern (1 to 20 W/min).

The incremental treadmill test will be performed to determine aerobic training load. The modified Balke protocol, according to the basal level of physical fitness (a total time increment between eight and 12 minutes).

The incremental shuttle walking test will be conducted according to the description of Singh et al.

The daily physical activity (DPA) will be assessed with an accelerometer for three days.

Blood sample for inflammatory markers measurements will be collected to analyze of IL-1 beta, IL-6, IL-8, IL-10, TNF-alpha, using Duo Set ELISA kits from R & D Systems according to manufacturer's instructions.

Muscle strength with one repetition maximum (1RM) will be performed at middle deltoid (MD), biceps brachial (BB) and quadriceps femoris (QF). The following movements will also be evaluated: shoulder abduction, elbow flexion and knee extension.

Patients are going to be randomized to pulmonary rehabilitation or conventional physiotherapy program as follow:

Pulmonary rehabilitation: 8 week, twice weekly exercise program with aerobic treadmill and lower limb strength training.

Conventional program: 8 week, twice weekly conventional program with: L'Expiration Lente Totale Glotte Ouverte en decubitus Latéral (Eltgol), autogenous drainage (AD) and shaker with duration of 30 minutes each.

Patients will be reassessed in 1 and 3 years, measuring maximal incremental cycle ergometer test, incremental treadmill test, incremental shuttle walking test, accelerometer and muscle strength. All tests will follow the same patterns as the first assesment. Adicionally, exacerbations, hospitalization and survival in each year will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and / or CT of bronchiectasis without cystic fibrosis
* Clinically stable (no change in symptoms of dyspnea, quantity and color of the secretion)
* Greater than 18 and / or oxygen dependent at home
* Medical Research Council MRC ≥ 1.

Exclusion Criteria:

* Smokers or smoking history> 10 pack / years,
* Cystic fibrosis (CF)
* Chronic obstructive pulmonary disease (COPD)
* Asthma
* Pulmonary fibrosis (PF)
* Musculoskeletal limitations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The change in exercise capacity in patients with bronchiectasis | Up to 36 months
  Exercise capacity is measured by maximal cardiopulmonary exercise test on a cycle ergometer. The protocol will be used in ramp.
Pulmonary Function | Up to 36 months
  For the cohort follow up, forced expiratory volume in the first second will be primary outcome
Exacerbations and Hospitalizations per year | Up to 36 months
  For the cohort follow up, the frequency of exacerbations and hospitalizations will be evaluated
Survival in months | Up to 36 months
  For the cohort follow up, the survival will be evaluated in months.

OTHER OUTCOMES:
Peripheral muscle function is measured by | Up to 36 months
  The maximal voluntary contraction in upper and lower limb was applied during the visits.

CONTACTS AND LOCATIONS:
Overall Officials: Anderson Alves de Camargo, master's, Principal Investigator — University of Nove de Julho; Rejane Agnelo Silva de Castro, Student, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

REFERENCES:
- [Derived] de Camargo AA, de Castro RAS, Vieira RP, Oliveira-Junior MC, Araujo AA, De Angelis K, Rached SZ, Athanazio RA, Stelmach R, Corso SD. Systemic Inflammation and Oxidative Stress in Adults with Bronchiectasis: Association with Clinical and Functional Features. Clinics (Sao Paulo). 2021 Apr 16;76:e2474. doi: 10.6061/clinics/2021/e2474. eCollection 2021. PMID 33886789